CLINICAL TRIAL: NCT01177384
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled, Double-Blind Clinical Trial to Evaluate the Safety and Efficacy of the Addition of Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet/Exercise Therapy and Acarbose Monotherapy
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of the Addition of Sitagliptin in Participants With Type 2 Diabetes Mellitus Receiving Acarbose Monotherapy (MK-0431-130)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-130; 2010_543 (Other: Merck Registration Number); CTRI/2011/10/002072 (Registry Identifier: CTRI)
Record Dates: First submitted 2010-06-30; First posted 2010-08-09 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Acarbose; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg daily (q.d.) + acarbose (continuing the current stable dose of at least 50 mg three times daily [t.i.d.])
  Interventions: Drug: Sitagliptin phosphate; Drug: Acarbose; Drug: Glimepiride
- Placebo (Placebo Comparator): Placebo q.d. + acarbose (continuing the current stable dose of at least 50 mg t.i.d.)
  Interventions: Drug: Comparator: Placebo; Drug: Acarbose; Drug: Glimepiride

INTERVENTIONS:
Drug: Sitagliptin phosphate — Sitagliptin, 100 mg tablet once daily, orally for 24 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Comparator: Placebo — Placebo, to match sitagliptin tablet, once daily, orally for 24 weeks
  Arms: Placebo
Drug: Acarbose — Acarbose 50 mg or 100 mg tablet, 3 times daily, orally (continuing on the stable dose established prior to screening) for 24 weeks
  Other Names: Precose
Drug: Glimepiride — Participants not meeting specific glycemic goals during the study will use glimepiride as rescue therapy. For countries where glimepiride is not available, participants will receive a sulfonylurea marketed in that country as rescue therapy.
  Other Names: Amaryl®; Glimy

SUMMARY:
This study will evaluate whether the addition of sitagliptin reduces hemoglobin A1C (A1C) more than the addition of placebo for participants with type 2 diabetes mellitus (T2DM) on a steady dose of acarbose. The primary hypothesis is that the addition of sitagliptin 100 mg once daily (q.d.) reduces A1C more than the addition of placebo in participants with T2DM with inadequate glycemic control on acarbose monotherapy.

DETAILED DESCRIPTION:
The study includes an 8-week antihyperglycemic agent (AHA) wash-off period* (which includes a 2-week single-blind placebo run-in period) followed by a 24-week double-blind treatment period. All participants will receive open-label acarbose at a minimum dose of 50 mg three times daily (t.i.d.) during the run-in and treatment periods.

*: Wash-off only applicable to patients who were on acarbose and another AHA.

ELIGIBILITY:
Inclusion Criteria:

* has T2DM and is on acarbose alone at a stable dose of at least 50 mg t.i.d.(three times a day) for at least 10 weeks or on acarbose at a stable dose of at least 50 mg t.i.d. (three times a day) for at least 10 weeks in combination with another antihyperglycemic agent (AHA)
* is at least 18 years of age (for participants in India: between 18 and 65 years of age)
* male or female who is unlikely to conceive (not of reproductive potential, or agrees to remain abstinent or use [or have partner use] acceptable birth control if of reproductive potential)

Exclusion Criteria:

* has a history of type 1 diabetes mellitus
* use of thiazolidinedione (TZD), dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists, or insulin
* has the following cardiovascular disorders: acute coronary syndrome; new or worsening symptoms of coronary heart disease; coronary artery intervention; stroke or transient ischemic neurological disorder
* has liver or kidney disease
* has cancer or any clinically significant disease or disorder as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2013-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Wang W, Ning G, Ma J, Liu X, Zheng S, Wu F, Xu L, O'Neill EA, Fujita KP, Engel SS, Kaufman KD, Shankar RR. A randomized clinical trial of the safety and efficacy of sitagliptin in patients with type 2 diabetes mellitus inadequately controlled by acarbose alone. Curr Med Res Opin. 2017 Apr;33(4):693-699. doi: 10.1080/03007995.2016.1277200. Epub 2017 Jan 25. PMID 28035868
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431-130&kw=0431-130&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants randomized population. The participant flow module includes the second sequential randomization of a participant in the placebo group. Data for the second sequential randomization were excluded from the efficacy and safety analyses and the reason for not completed was a protocol violation.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 191 | 190 (Includes the second randomization of a participant)
Completed | 177 | 164
Not Completed | 14 | 26
Not completed — Adverse Event | 6 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 4
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 5 | 12

BASELINE CHARACTERISTICS:
Population: All participants randomized population. The baseline characteristics module does not include the second sequential randomization of a participant in the placebo group. Data for the second sequential randomization were excluded from the efficacy and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 191 | 189 | 380
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (8.9) | 57.8 (9.5) | 57.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 92 | 186
  Male | 97 | 97 | 194
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] — Percent of glycosylated hemoglobin
  Percent | 8.09 (0.79) | 8.08 (0.90) | 8.08 (0.85)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 177.3 (37.5) | 177.5 (40.2) | 177.4 (38.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: A1C is measured as a percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent. Efficacy analyses treated data as missing after the initiation of rescue therapy.
Time Frame: Baseline and Week 24
Population: Full Analysis Set, all randomized participants except those who: failed to take at least 1 dose of study treatment, lacked all post-randomization data for the A1C subsequent to at least 1 dose of study treatment, or lacked baseline data for the A1C. Last observation carried forward (missing data approach).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 185 | 180
Percent | -0.76 [-0.93 to -0.59] | -0.14 [-0.32 to 0.03]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA — The ANCOVA model included terms for treatment and prior antihyperglycemic agent (AHA) therapy status (on acarbose monotherapy, or on acarbose in combination with other AHA(s)) and a covariate for baseline A1C; Difference in least squares mean = -0.62, 95% CI 2-sided [-0.79 to -0.44]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 FPG minus Week 0 FPG. Efficacy analyses treated data as missing after the initiation of rescue therapy.
Time Frame: Baseline and Week 24
Population: Full Analysis Set, all randomized participants except those who: failed to take at least 1 dose of study treatment, lacked all post-randomization data for the FPG subsequent to at least 1 dose of study treatment, or lacked baseline data for the FPG. Last observation carried forward (missing data approach).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 187 | 183
mg/dL | -17.9 [-25.3 to -10.5] | -3.5 [-11.1 to 4.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA — The ANCOVA model included terms for treatment and prior AHA therapy status (on acarbose monotherapy, or on acarbose in combination with other AHA(s)) and a covariate for baseline FPG; Difference in least squares mean = -14.4, 95% CI 2-sided [-21.8 to -7.0]

3. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Time Frame: Up to Week 24 + 14 Day Post-Study Follow-up
Population: All participants as treated population defined as all randomized participants who received at least one dose of study drug. Data were excluded after the initiation of rescue therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 191 | 189
Participants | 62 | 58

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 24 Weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 191 | 189
Participants | 5 | 2

ADVERSE EVENTS:
Description: All participants as treated population. Participants received rescue therapy if they met specific glycemic goals. Serious adverse events include events that occurred either before or after receiving rescue therapy. Other adverse events only include those AEs that occurred prior to a participant receiving rescue therapy.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 10/191 | 1/189
Other Adverse Events (participants affected / at risk) | 0/191 | 0/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=191) | Placebo (N=189)
Cardia flutter (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.